CLINICAL TRIAL: NCT04020016
Title: A Study of Nalbuphine Extended-release (NAL ER) Oral Tablets in Subjects With Impaired Hepatic Function Compared to Healthy Subjects and Exploratory Effect on Itch
Brief Title: Nalbuphine ER Effects of Liver Disease on Pharmacokinetics and Itch
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trevi Therapeutics (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 182018 (TR10)
Record Dates: First submitted 2019-05-30; First posted 2019-07-15 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Nalbuphine; Hepatic Impairment
Keywords: nalbuphine; Pharmacokinetic; hepatic impairment

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label PK and safety study of NAL ER in subjects with impaired liver function compared to healthy subjects. It will be performed in 2 parts:
  Part 1: single-ascending-dose (SAD) cohorts
  Part 2: multiple-ascending-dose (MAD) cohort
  In Part 1 (SAD)-Dose Cohorts 1-5: Each of the cohorts will be dosed sequentially starting with the lowest dose. The drug kinetics in the hepatic impairment subject population will be compared relative to the healthy subject population (Cohort 5).
  Part 2 (MAD) - Dose Cohort 6: 6-8 subjects with mild hepatic impairment and 6-8 subjects with moderate hepatic impairment In Part 2 of the study (MAD), subjects will receive multiple doses ascending from 27 mg up to 162 mg over 13 days of dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Single Ascending Dose (Experimental): Impaired liver function subjects and healthy liver subjects single ascending dosing up to 162 mg BID of Nalbuphine ER
  Interventions: Drug: Nalbuphine ER
- Part 2 Multiple Ascending Dose (Experimental): Impaired liver function subjects will receive multiple ascending dosing up to 162 mg BID of Nalbuphine ER
  Interventions: Drug: Nalbuphine ER -

INTERVENTIONS:
Drug: Nalbuphine ER — Cohort 1: 6-8 subjects will receive 1 dose of 27mg and observed for 4 days. Cohort 2: 6-7 subjects will receive 1 dose of 54 mg and observed for 4 days. Cohort 3: 6-7 subjects will receive 1 dose of 108 mg and observed for 4 days. Cohort 4: 6-8 subjects will receive 1 dose of 162 mg and observed for 4 days. Cohort 5: 6-8 healthy subjects will receive dosing of NAL ER and observed for 4 days.
  Other Names: NAL ER
  Arms: Part 1 Single Ascending Dose
Drug: Nalbuphine ER - — Cohort 6: • 6-8 subjects with mild hepatic impairment and 6-8 subjects with moderate hepatic impairment. Doses will be subsequently escalated for each subject starting at 27 mg on Day 1 to twice daily, 12 hours apart, 27 mg, 54 mg, 108 mg, and 162 mg over 13 days.
  Other Names: NAL ER
  Arms: Part 2 Multiple Ascending Dose

SUMMARY:
This research study will evaluate the effect of liver disease on the pharmacokinetics (the breakdown of the drug in the body) of parallel-group, multiple oral doses nalbuphine extended release (NAL ER), tablets in people with liver disease (mild, moderate and severe), compared to people with normal liver function. The study will also test the safety and tolerability of the NAL ER, when it is given to subjects with mild, moderate and severe liver disease, compared to subjects with normal liver function. This protocol will also study the effects of this drug on itching in liver disease subjects if they report some itching prior to taking part in this study.

DETAILED DESCRIPTION:
The study is a three-center study that will include both a single-ascending-dose (SAD) portion and a multiple-ascending dose (MAD) portion. The PK, safety, and tolerability of single ascending doses (SAD) of NAL ER (4 dose levels) will be evaluated in subjects with mild, moderate and severe hepatic impairment.

The purpose of the SAD will be to assess the safety and PK parameters of the given dose levels in hepatic impaired subjects relative to a selected healthy subject control population as part of the overall NAL ER development program. The SAD will also allow a better understanding of the safety, tolerability and expected steady state PK characteristics in mild and moderate hepatic impairment prior to undertaking safety and itch suppression efficacy studies in this patient population.

In the MAD portion of this study, PK assessment will be carried out at steady state at each respective dose level at steady state during the titration over 13 days up to the highest planned therapeutic dose of 162 mg. It is well documented, in clinical practice and the opiate literature, that gradually increasing the dose of drug with a structured titration can reduce the frequency and severity of the expected AEs associated with initiation of therapy. The NAL ER clinical program utilizes this type of structured titration strategy, starting with once per day dosing at the 27 mg dose of NAL ER, and increasing the dose in a stepwise manner over the next 13 days to the target investigational dose of 162 mg twice daily. Pharmacokinetic steady state is reached

ELIGIBILITY:
Inclusion Criteria:

For Subjects with Hepatic Impairment (Cohort 1 to 4 and Cohort 6)

* Male or female with stable hepatic impairment, non-smoker and/or light smoker.
* Clinical diagnosis of liver cirrhosis
* Stable for study participation based upon medical history, physical examination, vital signs, ECGs, and screening clinical laboratory evaluations

Inclusion Criteria:

For Healthy Subjects (Cohort 5):

* Male or female, non-smoker and/or light smoker (up to 5 cigarettes or equivalent/day),
* Healthy as defined by:

  1. Normal hepatic function
  2. The absence of clinically significant illness and surgery within 4 weeks prior to dosing.

Exclusion Criteria:

For Subjects with Hepatic Impairment (Cohort 1 to 4 and Cohort 6)

* Clinically significant unstable medical conditions
* Clinically significant abnormalities of laboratory, ECG, pulse oximetry, or clinical data that would preclude participation in the study.
* History of any illness that might confound the results of the study or pose an additional risk to the subject by participation in the study.

Exclusion Criteria

For Healthy Subjects (Cohort 5):

* Diagnosis of liver disease
* History of heart problems.
* History of significant alcohol abuse or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Individual and mean plasma concentrations verses time curves will be evaluated as a function of dose | Day -1 to 14
  The PK of NAL ER will be measured in hepatic impaired subjects steady state as a function of dose.
Incidence of Treatment-Emergent Adverse Events as assessed by Pulse Oximetry and Electrocardiogram (ECG) | Day -1 to 14
  Hepatic impaired subjects will be monitored for by pulse oximetry and ECG for Treatment-Emergent Adverse Events from dosing of NAL ER

SECONDARY OUTCOMES:
Worst Itch Numerical Rating Scale (WI-NRS) measurement tool for rating of itch severity in the hepatic impaired population | Day -1 to Day 16
  WI-NRS measure will be used to determine the severity of itch experienced by subjects with hepatic impairment (for Cohort 6 only) at screening. Subjects will be completing the two forms (the "Night-time Itch" and the "Daytime Itch") at the same time during the screening visit and the average will be taken to determine the baseline severity. The scale is a 0 to 10 rating scale with 10 being the most severe itch experienced and 0 being no itching experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sciascia, Study Director — Trevi Therapeutics, Inc.
Locations (3):
- United States (3):
  - 01, Miami, Florida
  - 02, Miami, Florida
  - 03, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No